CLINICAL TRIAL: NCT01780389
Title: Open-label Milnacipran for Persistent Knee Pain One Year After Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00017445; SAV-MD-08
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Knee Pain After Total Knee Arthroplasty; Osteoarthritis Pain
Keywords: Knee; Pain; Osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milnacipran (Experimental): Open-label flexibly dosed milnacipran
  Interventions: Drug: Open-label flexibly dosed milnacipran

INTERVENTIONS:
Drug: Open-label flexibly dosed milnacipran
  Other Names: Savella

SUMMARY:
The current study examines the effects of milnacipran in patients who have chronic persistent knee pain one year or longer after total knee arthroplasty (TKA) to evaluate for a pain-relieving effect.

DETAILED DESCRIPTION:
The current study proposes to collect pilot data on the utility of open-label milnacipran for the treatment of pain and other outcomes in this unfortunate group of patients with chronic persistent pain after TKA. Among marketed serotonin norepinephrine reuptake inhibitors (SNRIs), milnacipran has a unique property in that it blocks serotonin and norepinephrine reuptake equally. It is plausible that equipotent reuptake inhibition may confer greater analgesic benefit compared to other agents, and in preclinical animal models milnacipran has shown superior effects of ameliorating hyperalgesia and allodynia compared to some other antidepressant drugs. Additionally, milnacipran does not have inhibitory effects on cytochrome P (CYP) 450 enzymes, no binding affinity to neurotransmitter receptors liable to cause adverse events, and simple pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female adult outpatient age 18 or older at the time of consent.
2. Subject has chronic persistent pain 1 year after TKA without history of new injury, infection, or implant failure.
3. Subject has VAS > or = 40 mm at screen and baseline visits.
4. Subject has an understanding, ability and willingness to fully comply with study procedures and restrictions.
5. Subject has the ability to provide written, personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related procedures.

Exclusion Criteria:

1. Subjects unable to complete assessments due to language or cognitive impairment
2. Subjects with a history of bipolar disorder or psychosis as confirmed by the Mini International Neuropsychiatric Interview (MINI).
3. Subject currently has (or had a history within the last 6 months of) a drug dependence or substance abuse disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision (DSM-IV-TR) criteria (excluding nicotine).
4. Subjects who are currently considered a suicide risk, any subject who has previously made a suicide attempt or who has a prior history of or are currently demonstrating active suicidal ideation.
5. Subject has any clinically significant ECG or clinically significant laboratory abnormality (including a positive urine drug screen) at Screening.
6. Subject has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that in the Investigator's opinion would prohibit the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol.
7. Subjects who do not agree to use adequate and reliable contraception throughout the study.
8. Subject previously completed, discontinued or was withdrawn from this study.
9. Subject has taken an investigational drug or taken part in a clinical trial within 30 days prior to Screening.
10. Subjects treated with antidepressant medication within 4 weeks of screening visit (6 weeks for fluoxetine).
11. Subjects with known sensitivity to milnacipran.
12. Subjects with liver disease or reduced liver function
13. Subjects with obstructive uropathies
14. Subjects who consume alcohol in amounts viewed by the Investigator to be contraindicated
15. Subjects taking monoamine oxidase inhibitors
16. Subjects with uncontrolled narrow angle glaucoma
17. Subjects who are pregnant, may become pregnant, or who are nursing
18. Subjects with seizure disorders
19. Subjects with bleeding disorders or use of other medications that may cause bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davi M Marks, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Marks DM, Bolognesi MP. Open-label milnacipran for patients with persistent knee pain 1 year or longer after total knee arthroplasty: a pilot study. Prim Care Companion CNS Disord. 2013;15(4):PCC.12m01496. doi: 10.4088/PCC.12m01496. Epub 2013 Jul 11. PMID 24392250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Milnacipran
Started | 5
Completed | 4 (One patient discontinued due to adverse event.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 5 patients enrolled, 4 completed, 1 terminated due to adverse event.
Arm/Group | Milnacipran
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Visual Analogue Scale(VAS).
Description: The primary outcome is change in pain VAS from baseline to 12 weeks (baseline score minus 12 week or endpoint score; positive number reflects reduction in pain score). The effect size was calculated using the VAS scores measured on a scale of 0 to 100 mm:
  0= absence of pain or no pain noted 100 = worst imaginable pain/as bad as can be The higher the score the greater the over all pain intensity.
Time Frame: baseline and endpoint 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Milnacipran-Open Label: Open-label flexibly dosed milnacipran for 12 weeks. Twice-daily dosing will be used and the typical titration schedule will be as follows:
  Day 1 - 12.5 mg every morning Day 2-3 - 12.5 mg twice a day Day 4-7 - 25 mg twice a day Day 8-84 - 50 mg twice a day
  Taper:
  Day 85-88 - 25 mg twice a day Day 89-92 - 12.5 twice a day Day 93-96 - 12.5 mg every morning
Arm/Group | Milnacipran-Open Label
Number analyzed (Participants) | 5
units on a scale | 44 (1.8)

2. Secondary Outcome: Change in Knee Society Score (KSS).
Description: KSS measures subjective pain and objective function by joint physical exam. This secondary outcome was the change in Knee Society Score(KSS)from baseline through 12 weeks.
  KSS scores measured on a scale of 0 to 100 mm:
  0 = absence of pain or no pain noted 100= worst imaginable pain/as bad as can be The higher the score the greater the over all pain intensity.
Time Frame: between baseline and endpoint (12 weeks or early termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Milnacipran Open Label: Open-label flexibly dosed milnacipran
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 5
units on a scale | 1.37 (0.76) [0.76 to 1.37]

3. Secondary Outcome: Global Rating of Change
Time Frame: Endpoint (12 weeks or early termination)
Population: Data not collected.
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Total Score of Multidimensional Fatigue Inventory (MFI-20)
Description: Measures subjective fatigue.20-item self-report instrument consisting of five scales: General Fatigue, Physical Fatigue, Reduced Activity, Reduced Motivation, and Mental Fatigue.
  Each scale contains four items rated on a scale of one to 5 with the scale score of one having the anchor of entirely true and the scale score of 5 having the anchor of no, not true. The five scales were identified through factor analysis and are assumed to measure different aspects of fatigue. Lowest possible total score = 20 (absent fatigue) Highest possible total score = 100 (maximum fatigue) Total mean cumulative scores were reported
Time Frame: Baseline to endpoint (12 weeks or early termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 5
units on a scale | 0.46 (.30)

5. Secondary Outcome: Change in the Beck Depression Inventory (BDI-II)
Description: The secondary outcome measure is change in Beck Depression Inventory. The scale for this inventory is:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. The higher the score the degree of depression.
Time Frame: Baseline to endpoint (12 weeks or early termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 5
units on a scale | 0.49 (0.16) [0.16 to 0.49]

6. Secondary Outcome: Change in the Montgomery Asberg Depression Rating Scale
Description: Staff-rated assessment of depressive symptoms. Scale is as follows:
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: Between baseline and endpoint (12 weeks or early termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 5
units on a scale | 0.78 (0.23)

7. Secondary Outcome: Change in Total Score of State Trait Anxiety Inventory (STAI)
Description: Assessment of subjective symptoms of current anxiety and chronic anxiety. There are 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
  Lowest total score is 40 (absent anxiety) Highest total score is 160 (maximum anxiety) Total mean cumulative scores were reported.
Time Frame: baseline and endpoint (12 weeks or early termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 5
units on a scale | 0.69 (0.21)

8. Secondary Outcome: Change in Total Score of Short Form-36 (SF-36), Measuring Perceived Quality of Life
Description: Subjective measure of perceived quality of life.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.
  The eight sections are:
  * vitality,
  * physical functioning,
  * bodily pain,
  * general health perceptions,
  * physical role functioning,
  * emotional role functioning,
  * social role functioning,
  * mental health
  Scale:
  0= lowest quality of life 100= high quality of life Higher scores reflect higher quality of life. Total mean cumulative scores were reported.
Time Frame: baseline and endpoint (12 weeks or early termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran Open Label
Number analyzed (Participants) | 5
units on a scale | 1.16 (0.47)

ADVERSE EVENTS:
Time Frame: 12 weeks between baseline visit and week 12 visit.
Arm/Group | Milnacipran
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) — Spontaneously reported
Headache (General disorders) | 1 (1) — Spontaneously reported
constipation (Gastrointestinal disorders) | 1 (1) — Spontaneously reported
painful ejaculation (Nervous system disorders) | 1 (1) — Spontaneously reported

LIMITATIONS AND CAVEATS:
Limitations include this was a small open label pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No